CLINICAL TRIAL: NCT02036281
Title: A Phase 1 Study of Substance P-Saporin in Terminal Cancer Patients With Intractable Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 102013-010; NCT01875432 (obsolete NCT alias)
Record Dates: First submitted 2014-01-10; First posted 2014-01-15 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Terminally Ill; Histologically-confirmed Advanced Cancer; Pain, Intractable
Keywords: Terminally ill , histologically-confirmed advanced cancer; Pain unrelieved by opioids
MeSH Terms: conditions — Pain, Intractable | interventions — substance P-saporin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SP-SAP ARM (Experimental): The first subject will be enrolled in the 1-mcg SP-SAP cohort. A percutaneous intraspinal catheter will be placed at the L5-S1 interspace and the catheter advanced 4-5 cm into the intrathecal space under fluoroscopic guidance. To confirm location, CSF will be aspirated and radioopaque contrast dye injected. 1-mL study drug will be mixed with 1-mL patient CSF fluid and administered intrathecally via the catheter. The catheter will be flushed with 1 mL bolus of saline. Four hours after injection (+15 min), the catheter will be removed and the exit site treated with Neosporin ointment and sterilely dressed. Subjects will be monitored in the recovery room for 4 hours and in the hospital for 24 hours and discharged home. Patients only receive a single IT dose.
  Interventions: Drug: Substance P-Saporin

INTERVENTIONS:
Drug: Substance P-Saporin

SUMMARY:
The subjects will be treated with a single dose of SP-SAP. They will receive the study drug SP-SAP via a percutaneous intraspinal catheter, they will be monitored for 4 hours and required to stay in the hospital for 24 hours for precautionary care. Their vital signs will be monitored and recorded immediately following the injection. After the catheter has been removed, the following assessments will be made physical exam including motor and sensory functions, and electrocardiogram. A neurologist will be available for consultation as needed.

Beginning dose of SP-SAP will be 1 -mcg for the first cohort.

Subsequent single patient dose cohorts as 2, 4, 8, 16, 32, 64 and 90 mcg intrathecally (into the spine). SP-SAP will be accrued and treated after four weeks observation for toxicities between cohorts.

Study duration will be up to 6 months from the start of SP-SAP administration.

DETAILED DESCRIPTION:
Screening (-7 days to Day 0)

* Physical exam and medical history;
* Vital signs;
* Blood tests;
* Pain measurements (6 daily pain questionnaires for 7 days prior to receiving study drug);
* Urine tests;
* Pregnancy test;
* Electrocardiogram (EKG), a tracing of the electrical activity of the heart;
* Collection of demographic information (age, sex, ethnic origin);

Study Drug:

SP-SAP will be administered via a spinal injection. Depending on when the subject is enrolled in the study, the dose of SP-SAP will be between 1 and 90 micrograms of SP-SAP

Therapy:

Subject will arrive at the UTSW Eugene McDermott Center for Pain Management 2 hours prior to treatment. The following will take place:

* Physical exam;
* Pain measurements (6 pain questionnaires);
* EKG;
* The subject will have a catheter inserted into their spine and will receive the study drug intrathecally (into their spine). The catheter will remain in their spine for 4 hours. Less than 1 tablespoon of spinal fluid will be collected for research purposes; and
* They will remain in the University of Texas Southwestern Medical Center Hospital for 24 hours for observation as a precaution.

Follow-Up will occur weekly for 8 weeks and then monthly for 4 months as needed.

During these visits the following will take place:

* Physical exam (including sensory and motor skills) and medical history;
* Vital signs;
* Two tablespoons of blood will be drawn from your arm by needle stick for blood tests;
* Pain measurements (6 pain questionnaires);
* Urine tests; and
* Electrocardiogram (EKG), a tracing of the electrical activity of the heart.

The subject will be asked to keep a diary to record any nausea and vomiting as well as a medication log to record the pain medications and dosage that they take between visits.

Each visit will take approximately 2 hours to complete

4 Month Follow-Up Informational data on the level of pain, adverse events, and sensory and motor function will be collected for the remaining 4 months of the study or until time of death. This information may be collected via patient diary, office visit or telephone interview.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Signed informed consent
3. Terminally ill cancer patients with intractable chronic pain in the pelvis, lower abdomen, back, or spine. "Terminal" refers to ≤ six-month life expectancy. "Intractable" is defined as pain uncontrolled with medications or procedures.
4. Minimal expected survival time of one month
5. ECOG Performance status of 0 - 3
6. Able to verbally report pain
7. Able to indicate pain on a VAS
8. Able to perform motor/sensory tests
9. Able to undergo a 4-h intrathecal catheter placement
10. Other therapeutic and palliative options have been exhausted

Exclusion Criteria:

1. Concurrent therapy with an investigational agent
2. Concurrent radiation or chemotherapy
3. Pregnancy or failure to use effective contraception in fertile males or females, and breast-feeding females. For all female patients of child-bearing potential, a negative pregnancy test (serum or urine) within ten days before start of the study treatment must be obtained. Female patients must agree to use effective contraception, or must be surgically sterile, or must be postmenopausal. Acceptable forms of birth control are: spermicide with condom, diaphragm, or cervical cap, IUD-intrauterine device, birth control pills, or abstinence. The rhythm method or Plan B are not considered acceptable forms of birth control. Male patients must agree to use effective contraception or be surgically sterile.
4. Diagnosis of intractable chronic pain of the chest, head, neck or upper extremities.
5. Active infection or ulcer at the lumbar injection site
6. Inability to receive lumbar intrathecal injection because of other factors
7. Diagnosis of meningitis or encephalitis
8. Other severe, acute or chronic medical or psychiatric condition that may increase the risk associated with study participation or, in the judgment of the investigator, would make the patient inappropriate for the study
9. Comorbidities at particular risk (i.e., CNS, CNS metastases, hydrocephalus or coagulopathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-01; Primary Completion 2016-09-28 (Actual); Study Completion 2016-09-28 (Actual)

PRIMARY OUTCOMES:
Response Evaluation Criteria | 8 weeks
  The response criteria are based on achievement of a 20% reduction in chronic pain or opioid dose within eight weeks of treatment as assessed by at least two of the measured parameters: VAS "pain bothersomeness." VAS "pain intensity," ODI, SF-36, EQ-5D, BDI, and medication use log. Safe doses of opioids will be determined by referring physician and symptoms are refractory if at maximal safe dose of opioids (not associated with severe side effects), the VAS score remains elevated above 3.

SECONDARY OUTCOMES:
Safety Tolerability | 6 months
  Analyses will be performed for all subjects having received at least one dose of study drug. The study will use the CTCAE version 4.0 for reporting of non-hematologic adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Frankel, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - University of California, San Diego Mores Cancer Center, La Jolla, California
  - UT Southwestern Medical Center Simmons Comprehensive Cancer Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No